CLINICAL TRIAL: NCT00496041
Title: Belgian Prospective Multicentre Registry on the Performance of the Smart Stent in the Superficial Femoral Artery According to the New Tasc II-classification
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2007/208
Record Dates: First submitted 2007-07-03; First posted 2007-07-04 (Estimated); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Peripheral Vascular Disease
Keywords: Stenosis (> 75%) or occlusion of the superficial femoral artery
MeSH Terms: conditions — Peripheral Vascular Diseases; Constriction, Pathologic | interventions — Registries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Smart Stent in the Superficial Femoral Artery . (Experimental)
  Interventions: Procedure: Registry

INTERVENTIONS:
Procedure: Registry — A Registry will be used.

SUMMARY:
This is a Belgian prospective multicentre registry on the performance of the Smart stent in the superficial femoral artery according to the new tasc II-classification.

ELIGIBILITY:
Inclusion Criteria:

* Stenosis (> 75%) or occlusion of the superficial femoral artery (lesion up to 3 cm distal to Hunter's canal)
* New TASC (2007) A, B, or C lesions
* Vessel diameter between 4.5 and 6.5 cm
* Debilitating claudication or critical limb ischemia (Rutherford 2 to 5)
* At least 1 outflow vessel down to the ankle
* Signed informed consent
* > Age 50, life expectancy > 1 year
* Capable of concluding the necessary follow-up visits

Exclusion Criteria:

* Refusal to participate in the study
* Acute ischemia
* Inflow lesions > 50%, not successfully corrected before the procedure
* Combination with other treatment with the exception of treatment to improve the inflow

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2007-07 (Actual); Primary Completion 2008-12-31 (Actual); Study Completion 2008-12-31 (Actual)

PRIMARY OUTCOMES:
Patency as defined by absence of occlusion or >50% restenosis rate at the level the treated lesion as determined by duplex control. | 1 year

SECONDARY OUTCOMES:
Patency as defined by absence of occlusion, whether or not after additional intervention to maintain this patency (primary and secondary patency rate) | 1 year
Target lesion revascularisation rate as defined by the number of new revascularisations (endovascular or open) carried out due to restenosis at the level of the stented lesion | 1 year
Target vessel revascularisation rate as defined by the number of new revascularisations (endovascular or open) carried out due to restenosis or a new stenosis in the SFA. | 1 year
Limbs-salvage rate | 1 year
Clinical success rate defined on improvement in symptoms according to the Rutherford classification by a minimum of 1 class. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Frank Vermassen, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website of the University Hospital Ghent — http://www.uzgent.be